CLINICAL TRIAL: NCT03307902
Title: Intradermal Hepatitis B Vaccination With Imiquimod in Occult Hepatitis B Infection
Brief Title: ID HBV Vaccination With Imiquimod in OBI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UW 15-106
Record Dates: First submitted 2017-09-27; First posted 2017-10-12 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B
Keywords: Vaccination
MeSH Terms: conditions — Hepatitis B | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Imiquimod + ID HBVv (Experimental): topical imiquimod + intradermal hepatitis B vaccination
  Interventions: Biological: Imiquimod + ID HBVv
- Aqueous + ID HBVv (Active Comparator): topical aqueous + intradermal hepatitis B vaccination
  Interventions: Biological: Aqueous + ID HBVv
- Imiquimod + IM HBVv (Active Comparator): topical imiquimod + intramuscular hepatitis B vaccination
  Interventions: Biological: Imiquimod + IM HBVv

INTERVENTIONS:
Biological: Imiquimod + ID HBVv — Imiquimod ointment + intradermal 10μg Sci-B-Vac vaccine
  Arms: Imiquimod + ID HBVv
Biological: Aqueous + ID HBVv — Aqueous ointment + intradermal 10μg Sci-B-Vac vaccine
  Arms: Aqueous + ID HBVv
Biological: Imiquimod + IM HBVv — Imiquimod ointment + intramuscular 10μg Sci-B-Vac vaccine
  Arms: Imiquimod + IM HBVv

SUMMARY:
During the course of chronic hepatitis B infection, patients may undergo hepatitis B surface antigen (HBsAg) seroclearance, resulting in undetectable circulating HBsAg. With the advance of sensitive nucleic acid detection techniques, HBsAg-negative subjects with detectable HBV DNA in sera or liver tissues can be identified. Patients who have undetectable HBsAg and yet detectable HBV DNA in sera or liver tissues are defined as having occult HBV infection (OBI). OBI as a cause of liver disease in HBsAg-negative patients remains clinically important [1,2]. Studies conducted by our research group had demonstrated that patients with HBsAg seroclearance could still develop flare of hepatitis B, advanced liver diseases and HCC [3-6]. Prevention of these complications in OBI patients by conventional intramuscular hepatitis B vaccination (HBVv) remains elusive with poor amnestic anti-HBs response [7].

The objective of this prospective double-blind randomized controlled trial is to evaluate the effect and safety of topical treatment with imiquimod immediately before intradermal vaccination with Sci-B-Vac™ in patients with OBI. Our a priori hypothesis is that imiquimod pretreatment would improve immune responses to Sci-B-Vac™ further in OBI patients, resulting in HBsAb conversion. Thereby preventing subsequent complications including flare of hepatitis, cirrhosis and HCC in these patients.

DETAILED DESCRIPTION:
This randomized double-blind placebo-controlled trial will compare the safety, immunogenicity and clinical efficacy of Sci-B-Vac™ with topical ointment pretreatment among 5 groups. Group 1: Intradermal Sci-B-Vac™ with topical imiquimod ointment pretreatment; Group 2: Intradermal Sci-B-Vac™ with topical aqueous cream (placebo) pretreatment; Group 3: Intramuscular Sci-B-Vac™ with topical imiquimod ointment pretreatment.

Vaccination Regimen and Data Collection Enrolled patients will be randomized into 3 groups after written informed consent. Each patient will receive a 3 doses Sci-B-Vac™ regime at 0, 1 and 6 months. Group 1 will receive a total of 10μg intradermal HBsAg each time with topical imiquimod ointment pretreatment; Group 2 will receive a total of 10μg intradermal HBsAg each time with topical aqueous cream pretreatment. Group 3 will receive a total of 10μg intramuscular HBsAg each time with topical imiquimod ointment pretreatment.

The primary outcome measurement will be the seroprotection rate of the HBVv at 12 months after the first dose of vaccination and the secondary outcome measurements will include the seroconversion rate, the GMT fold increase and the safety of the intradermal Sci-B-Vac™ with topical imiquimod treatment at other time points.

ELIGIBILITY:
Inclusion Criteria:

* Subjects recruited have to be aged ≥27 years (born before the universal hepatitis B immunization program for newborns introduced in Hong Kong in 1988), with documentation of loss of HBsAg without anti-HBs production during follow-up of the chronic hepatitis B infection in our clinics in Queen Mary Hospital. These patients should have normal liver function tests.
* Subjects have to give written informed consent.
* Subjects must be available to complete the study and comply with study procedures.
* Subjects are willing to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

* Subjects with a history or any illness that might interfere with the results of the study or participation in the study may pose additional risk to the subjects.
* Subjects have a recent history (documented, confirmed or suspected) of a flu-like disease within a week of vaccination.
* Subjects have a known allergy to components of the study vaccine Sci-B-Vac™.
* Subjects have a positive urine or serum pregnancy test within 24 hours prior to vaccination, or women who are breastfeeding.
* Subjects have an active neoplastic disease or a history of any hematologic malignancy.
* Subjects have known chronic active hepatitis C (anti-HCV+ve), autoimmune hepatitis or cirrhosis.
* Subjects have known active human immunodeficiency virus infection (anti-HIV+ve).
* Subjects have known chronic liver disease due to primary biliary cirrhosis, metabolic or hereditary causes.
* Subjects have received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study.
* Subjects participate in another clinical study during the current study.
* Subjects have axillary temperature ≥38°C or oral temperature ≥38.5°C within 3 days of intended study vaccination
* Subjects have a history of alcohol or drug abuse in the last 5 years.
* Subjects have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate to HBV at 12 month | 12 month
  Percentage of recruited subjects with anti-HBs antibody titre >10mIU/mL

SECONDARY OUTCOMES:
Seroprotection rate to HBV at 1 month | 1 month
  Percentage of recruited subjects with anti-HBs antibody titre >10mIU/mL
Seroprotection rate to HBV at 6 month | 6 month
  Percentage of recruited subjects with anti-HBs antibody titre >10mIU/mL
GMT of anti-HBs at 1 month | 1 month
  Geometric mean titre of anti-HBs antibody at 1 month after vaccination
GMT of anti-HBs at 6 month | 6 month
  Geometric mean titre of anti-HBs antibody at 6 month after vaccination
GMT of anti-HBs at 12 month | 12 month
  Geometric mean titre of anti-HBs antibody at 12 month after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No